CLINICAL TRIAL: NCT04850157
Title: Tislelizumab Combined With Intensity Modulated Radiation Therapy（IMRT) Neoadjuvant Treatment for Resectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: Tislelizumab Combined With IMRT Neoadjuvant Treatment for Resectable Hepatocellular Carcinoma With PVTT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-187R-1
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab+IMRT (Experimental)
  Interventions: Drug: Tislelizumab; Radiation: IMRT

INTERVENTIONS:
Drug: Tislelizumab — 200mg, Q3W
Radiation: IMRT — 4 Gy* 5 Fx,5Fx/Week

SUMMARY:
Due to the biological characteristics and liver anatomical characteristics of liver cancer, liver cancer cells easily invade the vascular system, especially the portal venous system, forming portal vein tumor thrombus (PVTT) , and its incidence is reported to be 44.0% ~ 62.2%. Once PVTT occurs in patients with liver cancer, the disease develops rapidly, and intrahepatic and extrahepatic metastasis, portal hypertension, jaundice, and abdominal effusion can occur in a short time with an average survival time of 2.7 months. PVTT is one of the major adverse factors for the prognosis of liver cancer and occupies an important weight influence in the clinical staging system of liver cancer. In some hepatocellular carcinoma (HCC) patients with PVTT and selective resectability, surgery versus non-surgery can lead to better survival of patients.

A retrospective analysis showed that neoadjuvant radiotherapy can reduce the extent of invasion of PVTT and improve postoperative survival in some HCC patients. Another prospective study showed that neoadjuvant radiotherapy could significantly improve the overall survival of resectable liver cancer with PVTT, and neoadjuvant radiotherapy could improve the 2-year survival of patients from 9.4% to 27.4% 27.4%, with an effective response of 20.7%.

This study is a prospective, single-center, single-arm study to assess the efficacy and safety of neoadjuvant therapy with tislelizumab combined with IMRT for resectable liver cancer with PVTT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma
* Patients with at least one measurable lesion
* Resectable primary lesion, PVTTⅡ-Ⅲtype
* No previous treatment for hepatocellular carcinoma
* Eastern Cooperative Oncology Group(ECOG): Performance Status(PS)score 0-1
* Child-Pugh score A
* Expected survival ≥ 3 months
* Baseline blood routine and blood biochemical indicators should meet the following criteria:

hemoglobin ≥ 90 g/L, absolute neutrophil count ≥ 1.5 × 10 ^/L, platelet count ≥ 75 × 10 ^/L aspartate or alanine aminotransferase 5 times the upper limit of normal (ULN), alkaline phosphatase ≤ 2.5 times the ULN, serum albumin ≥ 30 g/L; serum creatinine 1.5 times the ULN; international normalized ratio (INR)) ≤ 2 or prothrombin time (PT) more than the upper limit of normal range ≤ 6 seconds

* Appropriate to participate in this trial as assessed by the investigator before entering the study
* Male and female subjects of childbearing potential must agree to use an effective method of contraception throughout the study
* Signed informed consent.

Exclusion Criteria:

* Imaging showed distant metastasis
* Previous treatment with other effective regimens (including surgery, radiotherapy, systemic therapy, etc.)
* Previous allergic reactions to the same kind of drugs
* Pregnant or lactating patients
* Active hepatitis B or C (hepatitis B: HBsAg positive and Hepatitis B (HBV )DNA ≥ 1*10^4 IU/ml; hepatitis C: hepatitis C virus (HCV) antibody and HCV RNA positive, requiring simultaneous antiviral therapy)
* Pericardial effusion, uncontrolled pleural effusion or clinically severe ascites at screening
* History of interstitial lung disease, pneumonitis, or uncontrolled systemic disease, including diabetes, hypertension, pulmonary fibrosis, acute lung disease
* Suffering from severe cardiovascular disease within 12 months before screening, such as symptomatic coronary heart disease,≥II congestive heart failure, uncontrolled arrhythmia, infarction, etc
* Any active immunodeficiency or autoimmune disease at screening and/or any history of immunodeficiency or autoimmune disease that may recur (such as hypothyroidism or hyperthyroidism, interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, etc.)
* Use of steroids or other systemic immunosuppressive therapy 14 days before enrollment; use of steroids or other systemic immunosuppressive therapy
* Patients with other previous malignancies that are not cured; Patients with other previous malignancies that are not cured
* Immunocompromised patients, such as immunocompromised patients, such as human immunodeficiency virus (HIV) positive; positive
* With uncontrollable psychosis; With uncontrollable psychosis
* Other factors make the investigators think it is inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival( RFS) | Up to 2 years
  Defined as the time from the date of surgery to the date of disease recurrence or death whichever occur first

SECONDARY OUTCOMES:
Resection rate (R0 resection rate) | Up to 2 years
  Defined as the proportion of patients undergoing radical resection to the total subjects (R0 resection rate)
Objective response rate (ORR) assessed by mRECIST | Up to 2 years
  Defined as the proportion of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Overall survival (OS) | Up to 2 years
  Defined as the time from the date of treatment start to the date of death or to the date of last follow-up for patients alive
Adverse Events (AEs) | Up to 2 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0; Surgical safety including Intraoperative blood loss，PHLF assessed by ISGLS（2012），Postoperative complications evaluated by modified Clavien-Dindo system.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided